CLINICAL TRIAL: NCT02031003
Title: Effect of an Infant Formula With High 2-Palmitic Vegetable Oil or an Identical Formula Supplemented With Oligofructose on Stool Composition and Stool Characteristics in Healthy Term Infants in Taiwan
Brief Title: Effect of Infant Formulas Containing a New Fat Blend or the New Fat Blend Plus Fiber in Healthy Term Infants
Acronym: 9055A1-2000
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3611001
Record Dates: First submitted 2013-12-23; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Bottle Feeding
MeSH Terms: conditions — Bottle Feeding | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Other): Standard infant formula
  Interventions: Dietary Supplement: Infant formula
- Experimental 1 (Experimental): Standard infant formula containing a new fat blend
  Interventions: Dietary Supplement: Infant formula
- Experimental 2 (Experimental): Standard infant formula containing a new fat blend and fiber
  Interventions: Dietary Supplement: Infant formula
- Human Milk (HM) (No Intervention): Non-randomized Human Milk group

INTERVENTIONS:
Dietary Supplement: Infant formula — Infant formula
  Arms: Control; Experimental 1; Experimental 2

SUMMARY:
* The primary objective of the study was to compare stool composition (stool soap and non-soap fatty acids, total fatty acids, minerals, and other stool constituents) of infants randomized to receive either standard formula, or 1 of 2 innovative formulas containing a new fat blend or the new fat blend plus fiber.
* The secondary objectives were to evaluate among the feeding groups, stool characteristics (stool consistency and frequency), GI tolerance assessed by the Infant Gastrointestinal Symptom Questionnaire (IGSQ), and urinary markers (F2-isoprostanes and 8-hydroxy-2'-deoxyguanosine [8-OHdG], and urine osmolality and specific gravity).
* The primary safety objective was to describe the frequency of adverse events (AEs) among the formula-fed (FF) groups.
* The secondary safety objective was to describe anthropometric measures (weight, length, and head circumference) among the feeding groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term (no less than 37 weeks and no greater than 42 weeks) singleton infants; between 25 days to 45 days post natal age (date of birth = Day 0) and weight for age ≥3rd and ≤97th percentiles according to Taiwan growth charts at the time of study entry.
* Human milk fed infants were exclusively consuming and tolerating HM and the mother must have made the decision to continue to exclusively breastfeed.
* Formula-fed infants were exclusively consuming and tolerating a cow's milk infant formula and parents/LAR must have previously made the decision to continue to exclusively formula feed.

Exclusion Criteria:

* Infants receiving any amount of supplemental HM with infant formula feeding or vice versa
* Family history of siblings with documented cow's milk protein intolerance/allergy
* Major congenital malformations, suspected or documented systemic or congenital infections, evidence systemic diseases

Ages: 25 Days to 45 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Stool Composition | Day 28
  Stool soap and non-soap fatty acids, total fatty acids, minerals, and other stool constituents

SECONDARY OUTCOMES:
Stool Consistency determined using a 3-day stool diary | Days 14 and 28
  Stool consistency data is collected using a 3-day stool diary completed by parents just prior to the Day 14 and Day 28 clinic visits. Average stool consistency scores are recorded on a validated 5-point scale (1 = Watery, 2 = Runny, 3 = Mushy Soft, 4 = Formed, 5 = Hard).
Stool frequency determined using a 3-day stool diary | Day 14 and 28
  Stool frequency data is collected using a 3-day stool diary completed by parents just prior to the Day 14 and Day 28 clinic visits. The average number of stools per day is determined for each consecutive 3-day period.
GI Tolerance | Baseline, Day 14 and Day 28
  GI tolerance assessed by the Infant Gastrointestinal Symptom Questionnaire (IGSQ)
Incidence of adverse events | From ICF signing until 14 days after last study feeding
Anthropometric measurements (weight, length and head circumference) | Baseline, Day 14 and Day 28
  Observed anthropometry measurements and derived z-scores will be determined and summarized by feeding group and by study visit.
Urine osmolality | Baseline and Day 28
  Measure of hydration status
Urine pH | Baseline and Day 28
  Measure of hydration status

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Chang Gung Medical Foundation - LinKuo Branch, Linkuo, Tao-Yuan County
  - Mackay Memorial Hospital - Hsinchu Branch, Hsinchu
  - Chang Gung Medical Foundation, Taipei Branch, Taipei
  - Mackay Memorial Hospital, Taipei

REFERENCES:
- [Derived] Nowacki J, Lee HC, Lien R, Cheng SW, Li ST, Yao M, Northington R, Jan I, Mutungi G. Stool fatty acid soaps, stool consistency and gastrointestinal tolerance in term infants fed infant formulas containing high sn-2 palmitate with or without oligofructose: a double-blind, randomized clinical trial. Nutr J. 2014 Nov 5;13:105. doi: 10.1186/1475-2891-13-105. PMID 25373935